CLINICAL TRIAL: NCT00364065
Title: A Randomized, Controlled, Double-Blind, Pilot Study to Evaluate Ferris PainWrap, a Semipermeable Hydrophilic Polymeric Membrane, in the Treatment of Chronic Low Back Pain
Brief Title: Study to Evaluate Ferris PainWrap in the Treatment of Chronic Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pain and Rehabilitation Medicine (Other)
Collaborators: Ferris Mfg. Corp. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00003008
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

INTERVENTIONS:
Device: Ferris PainWrap

SUMMARY:
The purpose of this study is to see if the Ferris PainWrap is effective in the treatment of chronic low back pain.

DETAILED DESCRIPTION:
This is a phase 4 study to determine if a semipermeable hydrophilic membrane marketed as Ferris PainWrap can relieve low back pain more effectively than a placebo wrap. In the United States, the prevalence of low back pain of at least 1 month's duration is about 15% and its incidence is 5%. It is one of the two most common pain complaints. Low back pain is thus a major health problem in this country and worldwide. Treatment that relieves low back pain and restores function would be of great benefit to the individual and the community at large, particularly if the treatment is convenient and has no significant adverse effects. Ferris PainWrap was originally developed as a burn dressing and is commercially available for this purpose. The Food and Drug Administration approved the material as Ferris Hydrophilic Dressing for marketing in interstate commerce prior to May 28, 1976, the enactment date of the Medical Device Amendments. The material is classified as a medical device. It was found to relieve pain, inflammation, swelling, and bruising over traumatized areas. Subsequently, it appeared to relieve low back pain in informal, open (non-blinded) trials. The proposed mechanism for low back pain relief is by alteration of cutaneous A-beta receptor and possibly cutaneous A-delta fiber function through shifts in sodium and water concentrations in the skin. This study will compare a "no dose" placebo to a "high-dose" back wrap. It is a one year pilot study which will be randomized, double-blinded, and controlled, comparing Ferris PainWrap to an identical appearing placebo back wrap in individuals with chronic low back pain of three months duration or longer.

ELIGIBILITY:
Inclusion Criteria:

* English speakers, necessary to understand the protocol and communicate observations to the investigators
* Low back pain of 3 months or longer. Acceptable conditions include non-specific low back pain or pain associated with lumbar spondylosis without neurological impairment associated with the stenosis.
* Numerical Pain Rating Scale value of 4.5 or higher, estimated for the past week where 0=no pain and 10=worst possible pain.
* Pain must interfere in some way with daily activities, assessed by Roland and Morris Disability Survey.
* Beck Depression Inventory score of 20 or less.
* Physical examination findings of tenderness, muscle spasm or taut bands, or myofascial trigger points in the low back region. The low back region is defined as the lumbosacral region, below the 12th thoracic vertebra down to the sacro-coccygeal junction, and extending laterally to the plane of the lumbar vertebral transverse processes.

Exclusion Criteria:

* Pregnancy
* NPR rating score of less than 4.5.
* Neurologic impairment in the legs (absent knee or ankle deep tendon reflexes, dermatome sensory loss or weakness) that indicates lumbar radiculopathy.
* Presence of cancer (previous diagnosis of cancer, or treated cancer with no sign of recurrence for 5 years is acceptable).
* Presence of systemic disease that can cause low back pain (endometriosis, prostatitis, chronic renal disease, recurrent urinary tract infections, or other acute infections, not including simple upper respiratory infections without significant coughing).
* Pending litigation involving back injury.
* Back related disability.
* Lumbar laminectomy.
* Subjects cannot have participated in other research studies within 3 months of starting this study.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-09; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Numerical pain rating scale

SECONDARY OUTCOMES:
Pain pressure threshold as determined by the Fischer algometer
Number of tender regions, taut bands, reproduction of usual and referred pain, recorded as present or absent
Range of motion as measured by inclinometer
Roland Morris Back Pain Disability score
Short Form-36 score
Daily count of analgesics taken
Pain diary, rating low back pain as none, mild, moderate, or severe

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Gerwin, MD, Principal Investigator — Assistant Professor, Johns Hopkins School of Medicine
Locations (1):
- Pain and Rehabilitation Medicine, Bethesda, Maryland, United States